CLINICAL TRIAL: NCT04513158
Title: Convalescent Plasma in the Early Treatment of High-Risk Patients With SARS-CoV-2 (COVID-19) Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Newly reported data at the time indicated that alternative therapies were more effective than CP for early treatment of high-risk patients with COVID-19.
Sponsor: Joseph M. Flynn, D.O., MPH (Other)
Responsible Party: Sponsor-Investigator, Joseph M. Flynn, D.O., MPH, Principal Investigator, Norton Healthcare
Organization: Norton Healthcare (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-N0124
Record Dates: First submitted 2020-08-06; First posted 2020-08-14 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Covid19
Keywords: SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: All hospitalized patients meeting study inclusion/exclusion criteria and providing informed consent for participation in the study will receive one unit (approximately 200 mL) of convalescent plasma over one hour to with data collection of routine physical exams/clinical assessments (daily) and routine lab results (every 3 days).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Study is single arm all patients hospitalized meeting inclusion/exclusion criteria and providing informed consent to receive one unit (approximately 200 mL) of convalescent plasma with data collected daily on routine (non-research) clinical assessments/physical exams and lab results.
  Interventions: Biological: Convalescent Plasma

INTERVENTIONS:
Biological: Convalescent Plasma — Plasma obtained from individuals previously diagnosed with SARS-CoV-2 (COVID-19) is administered to hospitalized patients meeting inclusion/exclusion criteria and have provided informed consent.

SUMMARY:
This study proposes to evaluate the therapeutic efficacy, immunologic effects and normalization of laboratory parameters for patients at high risk for mortality when infected by SARS-CoV-2 (COVID-19) when administered one unit (approximately 200 mL) of convalescent plasma administered over a period of one hour. Following administration of the convalescent plasma, physical exam/clinical assessment information is collected daily and routine lab result data is collected every three days.

DETAILED DESCRIPTION:
Following the administration of one unit (approximately 200 mL) of convalescent plasma over one hour, the study proposes to determine the therapeutic efficacy (response rate) of convalescent plasma infusion in patients at high risk for mortality when infected by SARS-CoV-2 (COVID-19) by prevention of progression to severe or life threatening COVID-19 during the current hospitalization as determined by evaluating if the patient experienced the following the following: respiratory rate >30/min, Blood oxygen saturation <93%, partial pressure of arterial oxygen to fraction of inspired oxygen ration <300, or received a medical diagnosis of respiratory failure, septic shock or multiple organ dysfunction/failure. This will be captured from the daily physical exam/clinical assessment done as part of routine care and at discharge.

The study also proposes to determine the immunologic effects of convalescent plasma infusion as measured by serial SARS-CoV-2 Ag levels through RT-PCR measured by CoV PCR collected at enrollment, day 7 and discharge.

Finally, the study intends to measure normalization of laboratory parameters for risk which will be documented every 3 days while the patient is hospitalized until the time that lab value returns to within the institution's normal range.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SARS-CoV-2 infection via RT-PCR or FDA approved testing.
* Patients must also have the following indications for enrollment:
* i. D-Dimer > 500 ng/ml FEU OR
* ii. IL-6> 5 pg/mL

With any of the following:

* iii. Lymphocytes < 0.8 103/ul OR
* iv. LDH > 700 U/L OR
* v. CK > 170 U/L OR
* vi. CRP > 1.0 mg/dl OR
* vii. Ferritin > 1000 ng/ml

AND one of the following:

* viii. Age over 60 years
* ix. Underlying Active Malignancy
* x. Cardiovascular Disease
* xi. Active Tobacco Use
* xii. History of Pulmonary Volume Reduction Surgery
* xiii. Hypertension
* Prior Treatment: Patients are still eligible for this trial if active antimicrobial agents are in use. Patients are also eligible if they had been treated on COVID-19 clinical trial in the course of their disease.
* Age ≥ 18 years.
* The effects of allogeneic plasma infusion on the developing fetus is unknown. For this reason women who are pregnant are not eligible to participate.
* Agrees to required laboratory data collected which will include the baseline organ function and regular ongoing assessments done as part of routine care.
* Ability to understand and the willingness to sign a written informed consent document or ability to have consent provided by Legally Authorized Representative.

Exclusion Criteria:

* 4.2.1 Patients who do not meet above inclusion criteria are not eligible.
* 4.2.2 Patients may not be receiving any other investigational agents.
* 4.2.3 History of allergic reactions attributed to previous transfusion history.
* 4.2.4 Respiratory rate >30/min
* 4.2.5 Blood oxygen saturation <93%
* 4.2.6 Partial pressure of arterial oxygen to fraction of inspired oxygen ration <300
* 4.2.7 Diagnosis of respiratory failure, septic shock or multiple organ dysfunction/failure

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Flynn, DO, MPH, Principal Investigator — Norton Healthcare
Locations (4):
- United States (4):
  - Norton Hospital, Louisville, Kentucky
  - Norton Women's and Children's Hospital, Louisville, Kentucky
  - Norton Audubon Hospital, Louisville, Kentucky
  - Norton Brownsboro Hospital, Louisville, Kentucky

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Bonow RO, Fonarow GC, O'Gara PT, Yancy CW. Association of Coronavirus Disease 2019 (COVID-19) With Myocardial Injury and Mortality. JAMA Cardiol. 2020 Jul 1;5(7):751-753. doi: 10.1001/jamacardio.2020.1105. No abstract available. PMID 32219362
- [Background] Rodriguez-Morales AJ, Cardona-Ospina JA, Gutierrez-Ocampo E, Villamizar-Pena R, Holguin-Rivera Y, Escalera-Antezana JP, Alvarado-Arnez LE, Bonilla-Aldana DK, Franco-Paredes C, Henao-Martinez AF, Paniz-Mondolfi A, Lagos-Grisales GJ, Ramirez-Vallejo E, Suarez JA, Zambrano LI, Villamil-Gomez WE, Balbin-Ramon GJ, Rabaan AA, Harapan H, Dhama K, Nishiura H, Kataoka H, Ahmad T, Sah R; Latin American Network of Coronavirus Disease 2019-COVID-19 Research (LANCOVID-19). Electronic address: https://www.lancovid.org. Clinical, laboratory and imaging features of COVID-19: A systematic review and meta-analysis. Travel Med Infect Dis. 2020 Mar-Apr;34:101623. doi: 10.1016/j.tmaid.2020.101623. Epub 2020 Mar 13. PMID 32179124
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] The Novel Coronavirus Pneumonia Emergency Response Epidemiology Team. The Epidemiological Characteristics of an Outbreak of 2019 Novel Coronavirus Diseases (COVID-19) - China, 2020. China CDC Wkly. 2020 Feb 21;2(8):113-122. No abstract available. PMID 34594836
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Zhao J, Yuan Q, Wang H, Liu W, Liao X, Su Y, Wang X, Yuan J, Li T, Li J, Qian S, Hong C, Wang F, Liu Y, Wang Z, He Q, Li Z, He B, Zhang T, Fu Y, Ge S, Liu L, Zhang J, Xia N, Zhang Z. Antibody Responses to SARS-CoV-2 in Patients With Novel Coronavirus Disease 2019. Clin Infect Dis. 2020 Nov 19;71(16):2027-2034. doi: 10.1093/cid/ciaa344. PMID 32221519
- [Background] Jean SS, Lee PI, Hsueh PR. Treatment options for COVID-19: The reality and challenges. J Microbiol Immunol Infect. 2020 Jun;53(3):436-443. doi: 10.1016/j.jmii.2020.03.034. Epub 2020 Apr 4. PMID 32307245
- [Background] Bhatraju PK, Ghassemieh BJ, Nichols M, Kim R, Jerome KR, Nalla AK, Greninger AL, Pipavath S, Wurfel MM, Evans L, Kritek PA, West TE, Luks A, Gerbino A, Dale CR, Goldman JD, O'Mahony S, Mikacenic C. Covid-19 in Critically Ill Patients in the Seattle Region - Case Series. N Engl J Med. 2020 May 21;382(21):2012-2022. doi: 10.1056/NEJMoa2004500. Epub 2020 Mar 30. PMID 32227758
- [Background] Baron SA, Devaux C, Colson P, Raoult D, Rolain JM. Teicoplanin: an alternative drug for the treatment of COVID-19? Int J Antimicrob Agents. 2020 Apr;55(4):105944. doi: 10.1016/j.ijantimicag.2020.105944. Epub 2020 Mar 13. PMID 32179150
- [Background] Mair-Jenkins J, Saavedra-Campos M, Baillie JK, Cleary P, Khaw FM, Lim WS, Makki S, Rooney KD, Nguyen-Van-Tam JS, Beck CR; Convalescent Plasma Study Group. The effectiveness of convalescent plasma and hyperimmune immunoglobulin for the treatment of severe acute respiratory infections of viral etiology: a systematic review and exploratory meta-analysis. J Infect Dis. 2015 Jan 1;211(1):80-90. doi: 10.1093/infdis/jiu396. Epub 2014 Jul 16. PMID 25030060
- [Background] Lim VW, Tudor Car L, Leo YS, Chen MI, Young B. Passive immune therapy and other immunomodulatory agents for the treatment of severe influenza: Systematic review and meta-analysis. Influenza Other Respir Viruses. 2020 Mar;14(2):226-236. doi: 10.1111/irv.12699. Epub 2019 Nov 16. PMID 31733048
- [Background] Cheng Y, Wong R, Soo YO, Wong WS, Lee CK, Ng MH, Chan P, Wong KC, Leung CB, Cheng G. Use of convalescent plasma therapy in SARS patients in Hong Kong. Eur J Clin Microbiol Infect Dis. 2005 Jan;24(1):44-6. doi: 10.1007/s10096-004-1271-9. PMID 15616839
- [Background] van Griensven J, Edwards T, de Lamballerie X, Semple MG, Gallian P, Baize S, Horby PW, Raoul H, Magassouba N, Antierens A, Lomas C, Faye O, Sall AA, Fransen K, Buyze J, Ravinetto R, Tiberghien P, Claeys Y, De Crop M, Lynen L, Bah EI, Smith PG, Delamou A, De Weggheleire A, Haba N; Ebola-Tx Consortium. Evaluation of Convalescent Plasma for Ebola Virus Disease in Guinea. N Engl J Med. 2016 Jan 7;374(1):33-42. doi: 10.1056/NEJMoa1511812. PMID 26735992
- [Background] Arabi Y, Balkhy H, Hajeer AH, Bouchama A, Hayden FG, Al-Omari A, Al-Hameed FM, Taha Y, Shindo N, Whitehead J, Merson L, AlJohani S, Al-Khairy K, Carson G, Luke TC, Hensley L, Al-Dawood A, Al-Qahtani S, Modjarrad K, Sadat M, Rohde G, Leport C, Fowler R. Feasibility, safety, clinical, and laboratory effects of convalescent plasma therapy for patients with Middle East respiratory syndrome coronavirus infection: a study protocol. Springerplus. 2015 Nov 19;4:709. doi: 10.1186/s40064-015-1490-9. eCollection 2015. PMID 26618098
- [Background] Zhou G, Zhao Q. Perspectives on therapeutic neutralizing antibodies against the Novel Coronavirus SARS-CoV-2. Int J Biol Sci. 2020 Mar 15;16(10):1718-1723. doi: 10.7150/ijbs.45123. eCollection 2020. PMID 32226289
- [Background] Casadevall A, Pirofski LA. The convalescent sera option for containing COVID-19. J Clin Invest. 2020 Apr 1;130(4):1545-1548. doi: 10.1172/JCI138003. No abstract available. PMID 32167489
- [Background] Hung IF, To KK, Lee CK, Lee KL, Chan K, Yan WW, Liu R, Watt CL, Chan WM, Lai KY, Koo CK, Buckley T, Chow FL, Wong KK, Chan HS, Ching CK, Tang BS, Lau CC, Li IW, Liu SH, Chan KH, Lin CK, Yuen KY. Convalescent plasma treatment reduced mortality in patients with severe pandemic influenza A (H1N1) 2009 virus infection. Clin Infect Dis. 2011 Feb 15;52(4):447-56. doi: 10.1093/cid/ciq106. Epub 2011 Jan 19. PMID 21248066
- [Background] Chen L, Xiong J, Bao L, Shi Y. Convalescent plasma as a potential therapy for COVID-19. Lancet Infect Dis. 2020 Apr;20(4):398-400. doi: 10.1016/S1473-3099(20)30141-9. Epub 2020 Feb 27. No abstract available. PMID 32113510
- [Background] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428
- [Background] Robeck J. Convalescent Plasma to Treat COVID-19. JAMA - J Am Med Assoc. 2020;Mar 27(Published online).
- [Background] Duan K, Liu B, Li C, Zhang H, Yu T, Qu J, Zhou M, Chen L, Meng S, Hu Y, Peng C, Yuan M, Huang J, Wang Z, Yu J, Gao X, Wang D, Yu X, Li L, Zhang J, Wu X, Li B, Xu Y, Chen W, Peng Y, Hu Y, Lin L, Liu X, Huang S, Zhou Z, Zhang L, Wang Y, Zhang Z, Deng K, Xia Z, Gong Q, Zhang W, Zheng X, Liu Y, Yang H, Zhou D, Yu D, Hou J, Shi Z, Chen S, Chen Z, Zhang X, Yang X. Effectiveness of convalescent plasma therapy in severe COVID-19 patients. Proc Natl Acad Sci U S A. 2020 Apr 28;117(17):9490-9496. doi: 10.1073/pnas.2004168117. Epub 2020 Apr 6. PMID 32253318
- [Background] Ruan Q, Yang K, Wang W, Jiang L, Song J. Clinical predictors of mortality due to COVID-19 based on an analysis of data of 150 patients from Wuhan, China. Intensive Care Med. 2020 May;46(5):846-848. doi: 10.1007/s00134-020-05991-x. Epub 2020 Mar 3. No abstract available. PMID 32125452
- [Background] Chen G, Wu D, Guo W, Cao Y, Huang D, Wang H, Wang T, Zhang X, Chen H, Yu H, Zhang X, Zhang M, Wu S, Song J, Chen T, Han M, Li S, Luo X, Zhao J, Ning Q. Clinical and immunological features of severe and moderate coronavirus disease 2019. J Clin Invest. 2020 May 1;130(5):2620-2629. doi: 10.1172/JCI137244. PMID 32217835
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Shi S, Qin M, Shen B, Cai Y, Liu T, Yang F, Gong W, Liu X, Liang J, Zhao Q, Huang H, Yang B, Huang C. Association of Cardiac Injury With Mortality in Hospitalized Patients With COVID-19 in Wuhan, China. JAMA Cardiol. 2020 Jul 1;5(7):802-810. doi: 10.1001/jamacardio.2020.0950. PMID 32211816
- [Background] Madjid M, Safavi-Naeini P, Solomon SD, Vardeny O. Potential Effects of Coronaviruses on the Cardiovascular System: A Review. JAMA Cardiol. 2020 Jul 1;5(7):831-840. doi: 10.1001/jamacardio.2020.1286. PMID 32219363
- [Background] Arentz M, Yim E, Klaff L, Lokhandwala S, Riedo FX, Chong M, Lee M. Characteristics and Outcomes of 21 Critically Ill Patients With COVID-19 in Washington State. JAMA. 2020 Apr 28;323(16):1612-1614. doi: 10.1001/jama.2020.4326. PMID 32191259
- [Background] Liu W, Tao ZW, Wang L, Yuan ML, Liu K, Zhou L, Wei S, Deng Y, Liu J, Liu HG, Yang M, Hu Y. Analysis of factors associated with disease outcomes in hospitalized patients with 2019 novel coronavirus disease. Chin Med J (Engl). 2020 May 5;133(9):1032-1038. doi: 10.1097/CM9.0000000000000775. PMID 32118640
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Gao Y, Li T, Han M, Li X, Wu D, Xu Y, Zhu Y, Liu Y, Wang X, Wang L. Diagnostic utility of clinical laboratory data determinations for patients with the severe COVID-19. J Med Virol. 2020 Jul;92(7):791-796. doi: 10.1002/jmv.25770. Epub 2020 Apr 10. PMID 32181911
- [Background] Liang W, Guan W, Chen R, Wang W, Li J, Xu K, Li C, Ai Q, Lu W, Liang H, Li S, He J. Cancer patients in SARS-CoV-2 infection: a nationwide analysis in China. Lancet Oncol. 2020 Mar;21(3):335-337. doi: 10.1016/S1470-2045(20)30096-6. Epub 2020 Feb 14. No abstract available. PMID 32066541
- [Background] Chan JW, Ng CK, Chan YH, Mok TY, Lee S, Chu SY, Law WL, Lee MP, Li PC. Short term outcome and risk factors for adverse clinical outcomes in adults with severe acute respiratory syndrome (SARS). Thorax. 2003 Aug;58(8):686-9. doi: 10.1136/thorax.58.8.686. PMID 12885985
- [Background] Tan L, Wang Q, Zhang D, Ding J, Huang Q, Tang YQ, Wang Q, Miao H. Lymphopenia predicts disease severity of COVID-19: a descriptive and predictive study. Signal Transduct Target Ther. 2020 Mar 27;5(1):33. doi: 10.1038/s41392-020-0148-4. No abstract available. PMID 32296069
- [Background] Tan L, Wang Q, Zhang D, Ding J, Huang Q, Tang YQ, Wang Q, Miao H. Correction: Lymphopenia predicts disease severity of COVID-19: a descriptive and predictive study. Signal Transduct Target Ther. 2020 Apr 29;5(1):61. doi: 10.1038/s41392-020-0159-1. eCollection 2020. PMID 32377400
- [Background] Zhang JJ, Dong X, Cao YY, Yuan YD, Yang YB, Yan YQ, Akdis CA, Gao YD. Clinical characteristics of 140 patients infected with SARS-CoV-2 in Wuhan, China. Allergy. 2020 Jul;75(7):1730-1741. doi: 10.1111/all.14238. Epub 2020 Feb 27. PMID 32077115
- [Background] Li B, Yang J, Zhao F, Zhi L, Wang X, Liu L, Bi Z, Zhao Y. Prevalence and impact of cardiovascular metabolic diseases on COVID-19 in China. Clin Res Cardiol. 2020 May;109(5):531-538. doi: 10.1007/s00392-020-01626-9. Epub 2020 Mar 11. PMID 32161990
- [Background] Zheng YY, Ma YT, Zhang JY, Xie X. COVID-19 and the cardiovascular system. Nat Rev Cardiol. 2020 May;17(5):259-260. doi: 10.1038/s41569-020-0360-5. PMID 32139904
- [Background] Emami A, Javanmardi F, Pirbonyeh N, Akbari A. Prevalence of Underlying Diseases in Hospitalized Patients with COVID-19: a Systematic Review and Meta-Analysis. Arch Acad Emerg Med. 2020 Mar 24;8(1):e35. eCollection 2020. PMID 32232218

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was open label, so there was no pre-assignment.
Period: Overall Study
Arm/Group | Treatment Arm
Started | 2
Completed | 1
Not Completed | 1
Not completed — Screen Failure | 1

BASELINE CHARACTERISTICS:
Population: Data was not collected or analyzed.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 0
Age, Categorical — Population: Data was not collected or analyzed.
Age, Continuous [unit: years] — Population: Data was not collected or analyzed.
Age, Customized — Population: Data was not collected or analyzed.
Sex/Gender, Customized — Population: Data was not collected or analyzed
  .
Sex: Female, Male — Population: Data was not collected or analyzed.
Ethnicity (NIH/OMB) — Population: Data was not collected or analyzed.
Race (NIH/OMB) — Population: Data was not collected or analyzed.
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Race/Ethnicity, Customized — Population: Data was not collected or analyzed.
Region of Enrollment [unit: participants] — Population: Data was not collected or analyzed.

OUTCOME MEASURES:

1. Primary Outcome: Determine the Therapeutic Efficacy (Response Rate) of Convalescent Plasma Infusion in Patients at High Risk for Mortality When Infected by SARS-CoV-2 (COVID-19).
Description: Measured by respiratory rate >30/min, blood oxygen saturation <93%, partial pressure of arterial oxygen to fraction of inspired oxygen ration <300 and received a medical diagnosis of respiratory failure, septic shock or multiple
Time Frame: Through study completion, an average of 30 days
Population: Data was not collected or analyzed.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 0

2. Secondary Outcome: Determine the Immunologic Effects of Convalescent Plasma Infusion
Description: SARS-CoV-2 Ag levels through RT-PCR
Time Frame: Through study completion, an average of 14 days
Population: Data was not collected or analyzed.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 0

3. Secondary Outcome: Absolute Lymphocyte Count (10*3/uL)
Description: Measure normalization of laboratory parameters for risk
Time Frame: Through study completion, an average of 14 days
Population: Data was not collected or analyzed.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 0

4. Secondary Outcome: Reatinine Kinase (mg/dL)
Description: Measure normalization of laboratory parameters for risk
Time Frame: Through study completion, an average of 14 days
Population: Data was not collected or analyzed.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 0

5. Secondary Outcome: C-reactive Protein (mg/dl)
Description: Measure normalization of laboratory parameters for risk
Time Frame: Through study completion, an average of 14 days
Population: Data was not collected or analyzed.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 0

6. Secondary Outcome: D-Dimer (ng/ml FEU)
Description: Measure normalization of laboratory parameters for risk
Time Frame: Through study completion, an average of 14 days
Population: Data was not collected or analyzed.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 0

7. Secondary Outcome: Interleukin-6 (pg/ml)
Description: Measure normalization of laboratory parameters for risk
Time Frame: Through study completion, an average of 14 days
Population: Data was not collected or analyzed.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 0

8. Secondary Outcome: Ferritin (ng/mL)
Description: Measure normalization of laboratory parameters for risk
Time Frame: Through study completion, an average of 14 days
Population: Data was not collected or analyzed.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Data was not collected or analyzed.
Description: Data was not collected or analyzed.
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Data was not collected or analyzed. Trial was stopped early because other therapy options became more readily available and the majority of room air patients were being discharged from the ED making finding eligible patients more difficult.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/58/NCT04513158/Prot_SAP_000.pdf